CLINICAL TRIAL: NCT02750384
Title: An Assessment of the Bioavailability and Effect of Food on DSM265 Granules in Healthy Adult Subjects
Brief Title: Bioavailability and Effect of Food on DSM265 Granules in Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategic decision based on preliminary results
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B16-963; MMV_DSM265_16_01 (Other Grant/Funding Number: The Medicines for Malaria Venture)
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers; Bioavailability
MeSH Terms: interventions — DSM265; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50% SDD granules, fasting (Experimental): 50% spray dried dispersion granules, fasting
  Interventions: Drug: DSM265 50% SDD granules
- 25% SDD powder for suspension, fasting (Active Comparator): 25% spray dried dispersion powder for suspension, fasting
  Interventions: Drug: DSM265 25% SDD powder for suspension
- 50% SDD granules, fed (Experimental): 50% spray dried dispersion granules, fed
  Interventions: Drug: DSM265 50% SDD granules

INTERVENTIONS:
Drug: DSM265 50% SDD granules — Single oral dose 400 mg
  Arms: 50% SDD granules, fasting; 50% SDD granules, fed
Drug: DSM265 25% SDD powder for suspension — Single oral dose 400 mg
  Arms: 25% SDD powder for suspension, fasting

SUMMARY:
This is a single-dose, fasting and non-fasting, open-label, randomized, three-regimen, parallel group study in 42 subjects

DETAILED DESCRIPTION:
This is a randomized, open label, single dose, parallel group study consisting of 3 groups of 14 subjects each. Subjects will be confined for 3 days followed by outpatient assessments until Day 21. Blood samples for assessment of DSM265 plasma concentrations will be collected for 480 hours after dosing.

This study will compare the relative bioavailability of the oral DSM265 50% spray dried dispersion (SDD) granules with that of a reference 25% SDD powder for suspension formulation, and evaluate the effect of food on the DSM265 50% SDD granules

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-child bearing potential:

  * surgically sterile (by hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy or bilateral tubal ligation) OR
  * postmenopausal (without use of hormonal contraceptive and spontaneous amenorrhea for 12 months and follicle stimulating hormone > 40 IU/mL age appropriate for menopause and no other medical explanation for amenorrhea)
* Males:

  * If he (including those who have had a vasectomy) is sexually active with female partner(s) of childbearing potential, he must agree, from Day 1 through 120 days after the dose of study drug to practice the continuous acceptable methods of contraception with his partner(s).
  * If he has a female partner who is postmenopausal or permanently sterile, the male subject must agree to use condoms from Day 1 through 120 days after the dose of study drug
* Females must have negative pregnancy tests:

  * at Screening within 28 days prior to initial study drug administration, and
  * prior to dosing on Study Day -1
* Body Mass Index at least 18.0 and less than / equal to 29.9. Body weight must be >50 kg
* General good health, based on medical history, physical examination, vital signs, laboratory profile and Electrocardiogram
* Voluntarily sign and date each informed consent, approved by an Institutional Review Board, prior to any screening or study procedures

Exclusion Criteria:

* Female who is pregnant, breastfeeding or is considering becoming pregnant during the study or for approximately 60 days after the dose of study drug
* Male who is considering fathering a child or donating sperm during the study or for 120 days after the last dose of study drug
* History of significant sensitivity to any drug
* History of epilepsy, any clinically significant cardiac, respiratory, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness
* History of gastric surgery (except phyloromoyotomy for pyloric stenosis during infancy), vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption
* Requirement for any over-the-counter or prescription medication, vitamins or herbal supplements, except contraceptives or hormone replacement therapy for females, on a regular basis
* Use of any medication, vitamins / herbal supplements except contraceptives or hormone replacement therapy for females, within 2 weeks prior to study drug administration or within 5 half-lives, whichever is longer
* Receipt of any drug by injection within 30 days or 5 half-lives, whichever is longer, prior to study drug administration, except parenteral hormonal contraceptives for females
* Receipt of any investigational product within 6 weeks prior to study drug administration or 5 half-lives, whichever is longer
* Recent (6-month) history of drug or alcohol abuse
* Consumption of alcohol within 72 hours prior to study drug administration
* Consumption of grapefruit or grapefruit products, Seville oranges, starfruit, or products containing any of these ingredients, and/or quinine/tonic water from 7 days prior to study drug administration
* Use of tobacco or nicotine-containing products within 6 months before study drug administration
* Positive for hepatitis A virus immunoglobulin M, hepatitis B surface antigen or hepatitis C virus antibody or HIV antibodies. Negative HIV status will be confirmed at Screening and results will be maintained confidentially
* Positive screen for drugs of abuse, or alcohol or cotinine or positive and clinically significant urine adulterants test
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product in 8 weeks prior to study drug administration
* Current enrollment in another clinical study
* Previous enrollment in this study
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive DSM265

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
DSM265 maximum observed plasma concentration (Cmax) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 time to Cmax (Tmax) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 observed concentration at 168 hours after dosing (C168) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 apparent terminal phase elimination rate constant (β) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 terminal elimination half-life (t1/2) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 area under the plasma concentration-time curve from time 0 to the time of the last measurable concentration (AUCt) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours
DSM265 area under the plasma concentration-time curve from time 0 to infinity (AUC∞) | Pre-dose and post-dose at 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168, 216, 312 and 480 hours

SECONDARY OUTCOMES:
safety evaluations | Pre-dose and Days 1, 2, 4, 6, 8, 10, 14, and 21
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: David, Carter, MD, Principal Investigator — AbbVie
Locations (1):
- AbbVie Clinical Pharmacology Research Unit (ACPRU), Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No